CLINICAL TRIAL: NCT02785328
Title: Sleep-dependent Memory Consolidation in Children With Sleep Diseases
Brief Title: Sleep and Memory in Children
Acronym: EnSOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL15_0226
Record Dates: First submitted 2016-05-20; First posted 2016-05-27 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Sleep Apnea; Temporo-central Epilepsy; Narcolepsy; High Intellectual Potential; Healthy Subject
Keywords: Memory; sleep; narcolepsy; apnea; epilepsy
MeSH Terms: conditions — Sleep Apnea Syndromes; Narcolepsy; Apnea; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- obstructive sleep apnoea (Experimental): The objective of this task is to evaluate the sleep-dependent consolidation abilities before and after treatment in children suffering from obstructive sleep apnoea syndrome.
  Interventions: Other: memory evaluation at V1 and V2 (with treatment)
- narcolepsy (Experimental): The objective of this task is to evaluate the sleep-dependent consolidation abilities before and after treatment in children suffering from narcolepsy.
  Interventions: Other: memory evaluation at V1 and V2 (with treatment)
- BECTS (Benign epilepsy with centro-temporal spikes) (Experimental): The objective of this task is to evaluate the sleep-dependent consolidation abilities before and after treatment in children suffering from BECTS.
  Interventions: Other: memory evaluation at V1 and V2 (with treatment)
- high intellectual potential (Experimental): The objective of this task is to evaluate the sleep-dependent consolidation abilities in children with high intellectual potential.
  Interventions: Other: memory evaluation at V1 (without treatment)
- healthy children (Experimental): The objective of this task is to evaluate the sleep-dependent consolidation abilities in healthy children.
  Interventions: Other: memory evaluation at V1 and V2 (without treatment)

INTERVENTIONS:
Other: memory evaluation at V1 and V2 (with treatment) — Overnight episodic and procedural memory consolidation performance will be assessed at V1 and V2. The performance will be correlated with sleep data, diurnal neuropsychological assessment and academic performance. The children receive drug treatment (BECTS and Narcolepsy) or surgical (OSA) as part of their routine care.
  Arms: BECTS (Benign epilepsy with centro-temporal spikes); narcolepsy; obstructive sleep apnoea
Other: memory evaluation at V1 (without treatment) — Overnight episodic and procedural memory consolidation performance will be assessed at V1. The performance will be correlated with sleep data, diurnal neuropsychological assessment and academic performance.
  Arms: high intellectual potential
Other: memory evaluation at V1 and V2 (without treatment) — Overnight episodic and procedural memory consolidation performance will be assessed at V1 and V2. The performance will be correlated with sleep data, diurnal neuropsychological assessment and academic performance.
  Arms: healthy children

SUMMARY:
Sleep exerts a dual effect on learning: on the one hand, good sleep quality allows good daytime aptitudes leading to knowledge acquisition. On the other hand, sleep after learning is necessary for knowledge consolidation. A key role of sleep has clearly been demonstrated in memory consolidation in adults. Sleep leads to strengthen memory by promoting brain plasticity. Surprisingly, sleep influence on learning stabilization has scarcely been studied during childhood and in children affected by sleep disorders. Yet, sleep disorders concern almost 30% of children and are frequently related to a worsening in academic performances. Classical neuropsychological evaluations of these children, based on daytime learning, often fail to determine cognitive profiles explaining their academic difficulties. The investigators hypothesize that a lack of sleep-dependent consolidation could take an active part in these children's cognitive and academic difficulties. This proposal aims at characterizing interactions between sleep, learning and memory processes that have not been studied in children of elementary school age (6-12 years). The investigators will evaluate sleep-dependent memory consolidation processes in children with sleep disorders before and after treatment and healthy controls. Neuropsychological testing and academic performances will be also evaluated.. The comparison of performances obtained before and after medical treatment, will allow to understand whether normalisation of sleep quality permits the restoration of sleep-dependent memory consolidation.

ELIGIBILITY:
Inclusion Criteria:

* aged between 6 and 12 y
* referred to the HFME for a suspicion of sleep apnea
* narcolepsy
* centro-temporal epilepsy
* high intellectual potential
* children without sleep disorders will be included in the healthy control group.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Memory performances | 6 months
  memory test : Björn Rasch, et al. (2007)
Memory performances | 6 months
  - Mirror drawing test : Nissen, et al. (2006).
Memory performances | 6 months
  - Word- pairs test : Urbain et al. (2011).
Memory performances | 6 months
  - Emotional memory test : Prehn-Kristensen et al. (2009).

SECONDARY OUTCOMES:
total sleep time (TST) | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
sleep efficiency (sleep time/time on bed) | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
sleep latency (time before sleeping after closing eyes) | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
number of awakenings | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
number of Stage 1 | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
number of Stage 2 | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
Slow-wave sleep (SWS) percentages | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
PS percentages | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
SWS time | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
PS latency (time between start of sleep and start of PS) | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
numbers of rapid eye movements | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
total cycle time (TCT) | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
TCT/TST ratio | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
WASO (wake after sleep onset) | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
apnoea/hypopnoea index | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
O2 desaturation | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
micro-arousal index | 3 months and 6 months
  standard full-night polysomnographic recording following the American Academy of Sleep Medicine recommendation will be performed at the hospital for the children suffering from sleep diseases (Morpheus, Medatec, Belgium) or at home for the healthy subjects (Dream, Medatec, Belgium). It will include electroencephalogram, electrooculogram, electromyogram, and electrocardiogram.
attention assessment | 3 months and 6 months
  Neuropsychological assessment will be standardized
short and long term memory | 3 months and 6 months
  Neuropsychological assessment will be standardized
executive functions | 3 months and 6 months
  Neuropsychological assessment will be standardized
depression and anxiety | 3 months and 6 months
  Neuropsychological assessment will be standardized
Intellectual Quotient | 3 months and 6 months
  Neuropsychological assessment will be standardized

CONTACTS AND LOCATIONS:
Overall Officials: Patricia FRANCO, MD PHD, Principal Investigator — Service d'exploration et pathologie du sommeil Hôpital Femme Mère Enfant, 59 bd Pinel 69677 BRON Cedex
Locations (1):
- Service d'exploration et pathologie du sommeil, Hôpital Femme Mère Enfant, 59 Bd Pinel, Lyon, Auvergne-Rhône-Alpes, France